CLINICAL TRIAL: NCT05193188
Title: A Multicenter Clinical Controlled Study of Anlotinib Combined With PD-1 Antibody on Unresectable High-grade Chondrosarcoma With Different IDH Genotypes
Brief Title: A Study of Anlotinib Combined With or Without PD-1 Antibody on Unresectable High-grade Chondrosarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LS2021-387
Record Dates: First submitted 2021-12-26; First posted 2022-01-14 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Chondrosarcoma
Keywords: Chondrosarcoma Anlotinib PD-1 monoclonal antibody
MeSH Terms: conditions — Chondrosarcoma | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib combined with PD-1 monoclonal antibody (Experimental): Anlotinib, a multi-target tyrosine kinase inhibitor，oral，12mg/10mg/8mg，2 weeks on and 1 week off; PD-1 monoclonal antibody，PD-1 inhibitor，Intravenous injection，once 3 week.
  Interventions: Drug: Anlotinib hydrochloride; Drug: PD-1 inhibitor
- Anlotinib monotherapy (Active Comparator): Anlotinib, a multi-target tyrosine kinase inhibitor，oral，12mg/10mg/8mg，2 weeks on and 1 week off.
  Interventions: Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Anlotinib hydrochloride — Anlotinib 12mg per person per day, continuous medication for 2 weeks and 1 week off, 3 weeks 1 cycle, until disease progression or intolerable toxicity
  Other Names: FuKeWei
Drug: PD-1 inhibitor — Intravenous injection, once every 3 weeks, until the disease progression or intolerable toxicity
  Arms: Anlotinib combined with PD-1 monoclonal antibody

SUMMARY:
There is no standard treatment for chondrosarcoma. Some small sample of studies has shown that anti-angiogenic TKIs show certain activity in the treatment of chondrosarcoma. PD-1 inhibitors, in recent years, have also been used in clinical practice and showed good efficacy. We intend to explore the response of chondrosarcoma to PD-1 monoclonal antibody and the influence of different IDH genotypes on PD-1 monoclonal antibody response.

DETAILED DESCRIPTION:
We intend to explore the response of chondrosarcoma to PD-1 monoclonal antibody and the influence of different IDH genotypes on PD-1 monoclonal antibody response. Patients with unresectable locally advanced or metastatic chondrosarcomas(CS), including high-grade (II-III) ordinary CS and dedifferentiated CS, are qualified. The experimental group was PD-1 monoclonal antibody combined with Anlotinib for treatment of unresectable locally advanced or metastatic CS, and the control group was anlotinib monotherapy. The treatment is continuous until the disease progression or intolerable toxicity. CS with disease progression in the control group was allowed to enter the experimental group to continue treatment. The primary endpoint was 6-month PFSR.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old, no gender limit; 2. ECOG PS score 0-2 points; 3. unresectable locally advanced or metastatic chondrosarcoma confirmed by histopathology, including high-grade (grade II-III) conventional CS and dedifferentiated CS; 4. Allow previous surgery, radiotherapy, or chemotherapy therapies; 5. Have at least 1 measurable lesion in accordance with the RECIST1.1; 6. The main organs are functioning normally and meet the following criteria within 7 days before treatment:

  * The standard of routine blood examination must be met (no blood transfusion and blood products within 14 days, no correction with G-CSF and other hematopoietic stimulating factors):

    1. Hemoglobin (HB) ≥90g/L;
    2. The absolute value of neutrophils (ANC) ≥ 1.5×109/L;
    3. Platelets (PLT) ≥100×109/L ② The biochemical inspection shall meet the following standards:

    <!-- -->

    1. Total bilirubin (TBIL)≤1.5×upper limit of normal (ULN);
    2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN, if there is liver metastasis, ALT and AST ≤ 5×ULN;
    3. Serum creatinine (Cr)≤1.5×ULN or creatinine clearance (CCr)≥60ml/min;

       ③ Urine protein <2+, and 24h urine protein quantitatively shows that the protein must be ≤ 1g;

       ④ Coagulation function: INR <2.0 and APTT≤1.5×ULN

       ⑤ Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (60%)

       ⑥ Thyroid function: TSH ≤ upper limit of normal (ULN); if abnormal, T3 and T4 levels should be considered, and T3 and T4 levels are normal and can be included in the group; 9. The fertile male or female agrees to use reliable contraceptive methods during treatment and at least 12 months after the last study drug is taken; 10. Sign the informed consent form with my consent, have good compliance and cooperate with follow-up.

       Exclusion Criteria:
* 1. Received anti-CTLA-4/PD-1/PD-L1 antibody treatment previously ; 2. Received anti-angiogenic TKI drugs (such as Anlotinib, Apatinib, Regofenib, etc.) or anti-angiogenic antibody drugs (such as Bevacizumab) previously; 3. Received other anti-tumor treatments within 4 weeks before enrollment, including systemic therapy, radiotherapy, major surgery, open biopsy, or participated in other clinical trials; 4. Patients who have not recovered from adverse events caused by any previous treatment to NCI-CTCAE (5.0) ≤1, excluding hair loss; 5. The investigator determines that there is a significant risk of bleeding, including but not limited to:

  1. Imaging shows that the tumor has invaded important blood vessels or it is judged by the investigator that the tumor is likely to invade important blood vessels and cause fatal hemorrhage during the follow-up study, or accompanied by large veins (iliac blood vessels, inferior vena cava, pulmonary vein, superior vena cava) tumor thrombus formation, or a history of aneurysm and the possibility of rupture;
  2. Received major surgical operations or had obvious traumatic injuries within 4 weeks before enrollment, or had any bleeding or bleeding event ≥ NCI-CTCAE Grade 3, or had any unhealed wounds, ulcers or fractures;
  3. There is a tendency for hereditary or acquired bleeding and thrombosis, such as hemophilia patients, blood coagulation dysfunction, thrombocytopenia, hypersplenism, etc.;
  4. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 ULN), have bleeding tendency, or are receiving thrombolytic or anticoagulant therapy;
  5. Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or similar drugs; Note: Under the premise that the international normalized ratio of prothrombin time (INR) ≤ 1.5, the use of low-dose heparin (daily dosage for adults is 6,000 to 12,000 U) or low-dose aspirin (daily dosage ≤100 mg); 6. The following symptoms or comorbidities exist:

  <!-- -->

  1. A history of hypertension, and can not be well controlled after treatment with 1-2 kinds of antihypertensive drugs (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg);
  2. Poorly controlled diabetes (fasting blood glucose> 10mmol/L);
  3. Significant cardiovascular damage includes, but is not limited to: unstable angina, myocardial ischemia or myocardial infarction, grade ≥2 congestive heart failure (New York Heart Association (NYHA) classification); occurred within 6 months Arterial/venous thrombotic events, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism;
  4. Sinus bradycardia of grade I or higher; or atrioventricular block of second degree or higher, or sinus arrest (except for pacemaker); arrhythmia (including QTc ≥480ms); need to take it at the same time to prolong the QTc interval Period drug
  5. Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral treatment;
  6. Urine routine test shows urine protein ≥ ++, and the 24-hour urine protein quantitative is confirmed to be> 1.0 g;
  7. Renal failure requires hemodialysis or peritoneal dialysis;
  8. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation, hematopoietic stem cell transplantation, or receiving systemic corticosteroids within 2 weeks before enrollment Or any other form of immunosuppressive therapy; Note: In the absence of active autoimmune diseases, inhaled or topical steroids and adrenal corticosteroids with a dose of> 10 mg/day prednisone equivalent dose are allowed, and the use of no more than 10 mg/day prednisone curative dose is allowed Adrenal corticosteroid replacement therapy, allowing glucocorticoids to be used as a preventive drug for hypersensitivity reactions (such as pre-docetaxel prophylaxis);
  9. Active or uncontrolled serious infection (≥CTC AE grade 2 infection) occurred within 4 weeks before enrollment;
  10. Judging by imaging studies, there is a central nervous system metastasis;
  11. Suffered from other malignant tumors in the past 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma, skin squamous cell carcinoma, and superficial bladder tumors;
  12. Those who have a history of psychotropic drug abuse and cannot be quit or have mental disorders;
  13. Those who have received ascites or pleural effusion drainage within 2 months of enrollment, or those who have uncontrollable pericardial effusion, pleural effusion and ascites;
  14. Complications of pulmonary fibrosis or interstitial pneumonia, or severe chronic obstructive pulmonary disease;
  15. Severe gastrointestinal diseases, such as gastric perforation, active peptic ulcer, etc.; 8. Combined medication

  <!-- -->

  1. During the study period, strong CYP3A inhibitors (such as itraconazole, telithromycin, clarithromycin, ritonavir, etc.) or moderate CYP3A inhibitors (such as ciprofloxacin) should be used;
  2. During the study period, strong CYP3A inducers (such as phenobarbital, phenytoin, rifampicin, carbamazepine) or moderate CYP3A inducers should be used;
  3. During the study period, it is necessary to take traditional Chinese medicines, especially those with anti-tumor activity; 9. Other

  <!-- -->

  1. It is expected that any form of systemic or local anti-tumor therapy will be taken during the study period;
  2. As judged by the investigator, there is a serious hazard to patient safety, concomitant diseases that may confuse the results of the study, or affect the patient to complete the study or any other conditions, such as a history of gastrointestinal disease that may affect the absorption of oral drugs.
  3. Those who have multiple factors that affect oral medications (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
  4. Allergic to the drugs in this study;
  5. Live vaccines have been vaccinated within 30 days before enrollment. Live vaccines include but are not limited to the following vaccines: measles, mumps, rubella, varicella/shingles (chickenpox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), typhoid vaccine.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
6month-PFSR | 6month
  Proportion of no disease progression after 6 months of medication

SECONDARY OUTCOMES:
ORR | 6month
  the proportion of patients with complete remission and partial remission
DCR | 6month
  the proportion of patients with complete remission, partial remission and stable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Binghao Li, Medical PhD, Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li B, Xie L, Liang J, Jiang Y, Wang K, Liu Y, Lin N, Huang X, Zhao K, Fan G, Liu M, Yan X, Qu H, Li H, Yang J, Zhou G, Ye Z. Anti-PD-1 antibody plus anlotinib vs. anlotinib alone in patients with refractory chondrosarcoma: A multicenter, non-randomized phase 2 FLAIL-C trial. Med. 2025 Nov 14;6(11):100809. doi: 10.1016/j.medj.2025.100809. Epub 2025 Aug 28. PMID 40882625